CLINICAL TRIAL: NCT01528579
Title: Effects of Different Exercise Programs for People With Chronic Whiplash Associated Disorders: a Prospective Randomized Study
Brief Title: Effects of Different Exercise Programs for People With Chronic Whiplash Associated Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Anneli Peolsson, Assoc Prof, PhD, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PeolssonAWADlong-term
Record Dates: First submitted 2012-01-22; First posted 2012-02-08 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Whiplash
Keywords: Whiplash; Rehabilitation; Physiotherapy; Exercises
MeSH Terms: conditions — Whiplash Injuries; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Neck Specific exercises (Active Comparator): Neck Specific exercises from a structured frame of exercises
  Interventions: Other: Neck Specific Exercises
- Behavioral approach (Active Comparator): Behavioral physiotherapeutic approach in combination with neck specific exercises from a structured well defined frame of exercises and how to treat the patient. 2 times a week for 3 months.
  Interventions: Behavioral: Behavioral approach combined with neck specific exercises
- Prescribed physical activity (Active Comparator): Prescribed physical activity from a physiotherapist without neck specific exercises
  Interventions: Other: Prescribed Physical activity

INTERVENTIONS:
Other: Neck Specific Exercises — 2 times a week for 3 months followed by encourages to continue on their own
  Arms: Neck Specific exercises
Behavioral: Behavioral approach combined with neck specific exercises — Behavioral physiotherapeutic approach combined with neck specific exercises 2 times a week for 3 months. Exercises will be chosen from a well defined and structured frame of exercises.
  Arms: Behavioral approach
Other: Prescribed Physical activity — Physical activity without neck specific exercises for 3 months
  Arms: Prescribed physical activity

SUMMARY:
Background:

Costs of health care consumption and sick leave 2006 in Sweden for Whiplash Associated Disorders (WAD) was estimated to be 4 billion Swedish crowns. Despite tremendous costs and personal sufferings there are only a few prospective randomized studies (RCT) in patients with chronic WAD, and none of them evaluating return to work, or the role of neck specific exercises with or without a combination of a behavioral approach compared with prescribed physical activity.

Aim:

The general aim of this RCT is to examine what neck-specific training with or without a combination with behavioral approach adds to prescribed physical activity of persons with chronic WAD with regard to pain intensity, physical and psychological function, health care consumption and return to work. Another aim is to study predictive factors of importance for a good outcome of rehabilitation.

Method:

After informed consent patients in age 18-63 years of age with WAD II-III with more than 6 months duration will be randomized to one out of the three alternatives of physiotherapy, treatment with medical exercise therapy with neck specific exercises (A),treatment with a behavioral approach combined with neck specific exercises (B), prescribed physical activity (C). Randomisation will be done by the central project leader. 200 patients will be included in the study. All physiotherapists engaged in the structured and well described treatment will be introduced in the program by the project leader. The measurements with good clinometric properties will be performed before treatment, after 12 weeks, 6, 12 and 24 months after inclusion into the study. Clinical measurements will be performed by a blinded investigator. Background data, disease-specific and generic data will be measured by self-evaluated answered questionnaires by the patients. Days of sick-leave will be collected from the Social Insurance Agency. Main outcomes of the measurements are pain intensity, neck specific disability and return to work. Cost-effectiveness will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-63 years
* WAD II-III
* Remaining problems (>10mm on 100mm Visual Analogue Scale (VAS) or >20% on Neck Disability Index (NDI) or at least moderate pin on NDI) at least 6 months but no more than 3 years after whiplash trauma

Exclusion Criteria:

* Myelopathy
* Earlier fracture or luxation of the cervical column, earlier neck injury
* Spinal tumour
* Spinal infection
* Surgery in the cervical column
* Malignity
* Systematic disease or another injury contraindicated to perform the treatment program or the measurements.
* Diagnosed severe psychiatric disorder
* Unconscious in connection to the trauma
* Known drug abuse
* Lack of familiarity with the Swedish language

Ages: 18 Years to 63 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 216 (Actual)
Dates: Start 2011-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Neck Disability Index (NDI) | Baseline and change after 3 and 6 months of exercises, 3 month, 6 month, 12 month and 24 month follow-up. Change from baseline to follow-ups. Twelve month follow-up is the most important follow-up to investigate change over time from baseline.
  NDI will be measured at baseline before intervention. Change from baseline in NDI will be measured at 3,6,12,and 24 months to investigate change over time. Baseline and change after three and six months of exercises and to investigate if a potential change of the exercises remain at 12 month and 24 month from baseline.

SECONDARY OUTCOMES:
Pain intensity on VAS | before intervention, 3, 6, 12 and 24 months follow-up. The outcome measure is going to report a change over time.
  Pain intensity is measured on a 100mm Visual Analogue Scale (VAS).
Pain Disability Index | before intervention, 3,6, 12, and 24 months follow-ups. The outcome measure is going to report a change over time.
Neck muscle endurance in seconds | before intervention, 3,6, 12, and 24 months follow-ups. The outcome measure is going to report a change over time.
Self-efficacy scale | before intervention, 3,6, 12, and 24 months follow-ups. The outcome measure is going to report a change over time.
Work Ability Index | before intervention and at 3, 6, 12 months and 24 months follow-up. The outcome measure is going to report a change over time.
Euroquol | before intervention, 3,6, 12, and 24 months follow-ups. The outcome measure is going to report a change over time.
SF-36 | before intervention, 3,6, 12, and 24 months follow-ups. The outcome measure is going to report a change over time.
Pain Catastrophizing Scale | before intervention, 3,6, 12, and 24 months follow-ups. The outcome measure is going to report a change over time.
Tampa Scale 11, short version | before intervention, 6, 12, and 24 months follow-ups. The outcome measure is going to report a change over time.
Neurological status | before intervention, 3,6, 12, and 24 months follow-ups. The outcome measure is going to report a change over time.
  Sensibility, reflexes,motor function upper extremeties, nerve tension test median nerve.
Pain drawing | before intervention, 3,6, 12, and 24 months follow-ups. The outcome measure is going to report a change over time.
  For the pain-drawing task, patients indicated the extent and the distribution of their pain on outlines of full front and back views of a human body. After the patients completed each pain-drawing, the distributions of symptoms will be coded on a seven-point scale (were 0 is no pain, and 6 is pain distributed in the hand), and where the pain was located in the cervical, thoracic, and/or the lumbar spine, in the front and the back of the body, will be indicated using a clear overlay template.
Clinical objective measures | before intervention, 3,6, 12, and 24 months follow-ups. The outcome measure is going to report a change over time.
  Range of motion of the neck and cervical kinesthesia (ability to reproduce the neutral head position from 30° cervical rotation with the eyes closed) will be measured with Cervical range of motion device (CROM).
  Balance (Static:sharpened Romberg's position with eyes closed. Dynamic: Walking in a figure-of-eight). Hand strength measured with a Jamar dynamometer. Dorsal and ventral eck muscle endurance measured in seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Anneli Peolsson, PhD, RPT, Study Chair — Linkoeping University
Locations (2):
- Sweden (2):
  - Linköping University, Linköping, Östergötland County
  - Department of Medical and Health Sciences, physiotherapy, Linköping, Östergötland County

REFERENCES:
- [Derived] Liew BXW, Scutari M, Peolsson A, Peterson G, Ludvigsson ML, Falla D. Investigating the Causal Mechanisms of Symptom Recovery in Chronic Whiplash-associated Disorders Using Bayesian Networks. Clin J Pain. 2019 Aug;35(8):647-655. doi: 10.1097/AJP.0000000000000728. PMID 31169550
- [Derived] Landen Ludvigsson M, Peterson G, Peolsson A. The effect of three exercise approaches on health-related quality of life, and factors associated with its improvement in chronic whiplash-associated disorders: analysis of a randomized controlled trial. Qual Life Res. 2019 Feb;28(2):357-368. doi: 10.1007/s11136-018-2004-3. Epub 2018 Sep 17. PMID 30225786
- [Derived] Ardern CL, Peterson G, Ludvigsson ML, Peolsson A. Satisfaction With the Outcome of Physical Therapist-Prescribed Exercise in Chronic Whiplash-Associated Disorders: Secondary Analysis of a Randomized Clinical Trial. J Orthop Sports Phys Ther. 2016 Aug;46(8):640-9. doi: 10.2519/jospt.2016.6136. Epub 2016 Jul 3. PMID 27374016
- [Derived] Ludvigsson ML, Peterson G, Dedering A, Falla D, Peolsson A. Factors associated with pain and disability reduction following exercise interventions in chronic whiplash. Eur J Pain. 2016 Feb;20(2):307-15. doi: 10.1002/ejp.729. Epub 2015 May 29. PMID 26031995
- [Derived] Peolsson A, Landen Ludvigsson M, Overmeer T, Dedering A, Bernfort L, Johansson G, Kammerlind AS, Peterson G. Effects of neck-specific exercise with or without a behavioural approach in addition to prescribed physical activity for individuals with chronic whiplash-associated disorders: a prospective randomised study. BMC Musculoskelet Disord. 2013 Oct 30;14:311. doi: 10.1186/1471-2474-14-311. PMID 24171699